CLINICAL TRIAL: NCT00067353
Title: Fluoride Varnish Trial in High Caries Preschoolers
Brief Title: Yakima Head Start Fluoride Varnish Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); The Yakima Valley Farm Workers Clinic (Other); Enterprise for Progress in the Community (Other); Washington State Migrant Council (Other)
Responsible Party: Philip Weinstein, DDS, Enterprise for Progress in the Community (EPIC) Head Start sites
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDCR-14403; R01DE014403 (NIH)
Record Dates: First submitted 2003-08-15; First posted 2003-08-19 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Dental Caries
Keywords: Early Childhood Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fluoride varnish

SUMMARY:
The aim of this study is to determine whether an annual application of three (3) fluoride varnish doses over two weeks is at least as effective in reducing cavities as the current semi-annual application.

DETAILED DESCRIPTION:
The study population will consist of pre-school aged children who are residents of Yakima County, in central Washington State. Children will be recruited from non-migrant Head Start programs for ethnic minority farmworker children in the Yakima Valley.

This study will be a randomized, double blinded trial with one experimental and one standard treatment group. Each participant will be randomly assigned to one of two study groups. The participant and the personnel conducting the study will not know to which study group the participant was assigned.

This trial has two study groups:

1. Massive Dose (Experimental):

   Annually for three years, children in the experimental group will receive three .30ml applications of 50mg NaF/mL fluoride varnish (CavityShieldÒ, Omni), followed 6 months later by three .30ml applications of placebo varnish in two weeks. There are 18 visits over the entire duration of the study. Each participant will receive a dental exam annually.
2. Semiannual Dose (Standard):

Annually for three years, children in the standard treatment group will receive one .30ml application of 50mg NaF/mL fluoride varnish (CavityShieldÒ, Omni) and two .30ml applications of placebo varnish in two weeks. They will receive this regimen again 6 months later. There are 18 visits over the entire duration of the study. Each participant will receive a dental exam annually.

Both the experimental and standard treatment children will receive basic restorative dental care on decayed surfaces only, as well as toothbrushes for the duration of the study period. Parents will fill out questionnaires about behaviors such as diet, hygiene and prior dental care. Results will inform future treatment regimens for high-caries-risk populations.

ELIGIBILITY:
Inclusion Criteria:

* Age 36-71 months
* Enrolled in participating Head Start Center
* Plan to stay in Yakima County for duration of the study
* One sound tooth surface present

Exclusion Criteria:

* No teeth present
* Developmentally unable to give oral assent

Ages: 36 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500
Dates: Start 2003-11; Primary Completion 2005-07 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Number of decayed, missing, or filled surfaces

CONTACTS AND LOCATIONS:
Overall Officials: Philip Weinstein, DDS, Principal Investigator — Washington State Head Start Sites
Locations (2):
- United States (2):
  - Enterprise for Progress in the Community (EPIC) Head Start sites, Lower Valley, Yakima County, Washington
  - Washington State Migrant Council Head Start sites, Lower Valley, Yakima County, Washington

REFERENCES:
- [Derived] Weinstein P, Spiekerman C, Milgrom P. Randomized equivalence trial of intensive and semiannual applications of fluoride varnish in the primary dentition. Caries Res. 2009;43(6):484-90. doi: 10.1159/000264686. Epub 2009 Dec 10. PMID 20016179